CLINICAL TRIAL: NCT00661830
Title: A Randomized, Double-blind, Multicenter Phase II Trial With Gemcitabine Plus Sorafenib Versus Gemcitabine Plus Placebo in Patients With Chemo-naive Advanced or Metastatic Adenocarcinoma of the Biliary Tract
Brief Title: Gemcitabine and Sorafenib in Advanced Biliary Tract Cancer (GEMSO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PD Dr Markus Möhler (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); Interdisciplinary Center for Clinical Trials (IZKS) (Unknown)
Responsible Party: Sponsor-Investigator, PD Dr Markus Möhler, MD, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC-GEMSO-2007
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-09

CONDITIONS: Adenocarcinoma
Keywords: advanced; metastatic; biliary; tract
MeSH Terms: conditions — Adenocarcinoma; Neoplasm Metastasis | interventions — Gemcitabine; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Gemcitabine + Sorafenib
  Interventions: Drug: Gemcitabine; Drug: Sorafenib
- 2 (Placebo Comparator): Gemcitabine + Placebo
  Interventions: Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 body surface i.v. first cycle at day 1, 8, 15, 22, 29, 36, 43. Next cycles at day 1, 8, 15.
Drug: Placebo — Placebo
  Arms: 2
Drug: Sorafenib — Sorafenib 400 mg bid orally continuously
  Arms: 1

SUMMARY:
This trial will be conducted to evaluate the efficacy, safety and tolerability of a combination of gemcitabine plus sorafenib in comparison of gemcitabine plus placebo as a first-line palliative therapy in chemo-naive advanced or metastatic CCC. There is strong scientific rationale for exploring the role of sorafenib in combination with gemcitabine in advanced CCC.

Sorafenib is a novel signal transduction inhibitor that prevents tumor cell proliferation and angiogenesis through blockade of the Raf/MEK/ERK pathway at the level of Raf kinase and the receptor tyrosine kinases VEGF-R2, R3 and PDGFR-β.

Mutations in these signaling pathways display by far the most common genetic alterations in CCC and overexpression correlates to poor prognosis. Furthermore, there is no evidence of a consistent or meaningful pharmacokinetic interaction between sorafenib and gemcitabine, suggesting that sorafenib can safely be combined with gemcitabine.

Clinical results of a combination of sorafenib and gemcitabine in a phase I study in pancreatic cancer suggested a therapeutic effect, and the safety and efficacy results together with the knowledge of the molecular pathology of CCC provide a rationale for a randomized, placebo-controlled phase II trial consisting of gemcitabine plus sorafenib in advanced CCC.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years and older
* Signed and dated informed consent before the start of specific protocol procedures
* Adenocarcinoma of the gallbladder or intrahepatic bile ducts or histologically proven hepatic metastases of an earlier resected and histologically proven biliary tract cancer

  * Not amenable to curative surgical resection
  * With at least one unidimensionally measurable target lesion in non-irradiated (or treated by photodynamic therapy, PDT) area (largest diameter ≥ 1 cm (spiral CT scan or MRI) or ≥ 2 cm (conventional CT scan)
  * With pain and biliary obstruction controlled
  * Cytologically or histologically confirmed
* Note : in case of uncertain biliary tract origin (e.g., intrahepatic CCCs), inclusion is possible if

  * extensive search for primary tumor (thoracic and abdomino pelvic CT scan, colonoscopy, upper digestive endoscopy, serum PSA level for men or mammography for women, and FDG-PET if possible) is negative
  * histological examination is consistent with bile duct adenocarcinoma, with IHC positive for cytokeratin 7 and 19 and negative for cytokeratin 20 [Shimonishi, 2000].
  * No histological evidence of hepatocellular carcinoma (HCC)
  * No prior palliative (radio)-chemotherapy (gemcitabine or fluoropyrimidine-based chemotherapy)
* Note:

  * previous adjuvant chemotherapy is allowed (completed since ≥ 6 months if containing gemcitabine or platinum salts);
  * previous irradiation (external radiotherapy, brachytherapy, chemoembolization) and PDT are allowed, provided that there is at least one unidimensionally measurable target lesion in untreated area
* Resolution of all side effects of prior surgical procedures to grade ≤ 1 (except for the laboratory values specified below)
* At least 4 weeks from any major surgery (at first dose of study drug)
* ECOG Performance Status of 0-2

Exclusion Criteria:

* Surgery (except diagnostic biopsy), external radiotherapy, brachytherapy, or PDT within 30 days prior to start of treatment.
* Other tumor type than adenocarcinoma (e.g. leiomyosarcoma, lymphoma) or a second cancer except in patients with squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix which has been effectively treated. Patients curatively treated and disease free for at least 5 years will be discussed with the sponsor before inclusion
* History of cardiac disease: congestive heart failure > NYHA class 2; active CAD (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
* Any of the following within the 12 months prior to starting the study treatment,: coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Ongoing cardiac dysrhythmias of grade ≥ 2, atrial fibrillation of any grade, or QTc interval > 450 msec for males or > 470 msec for females
* Hypertension that cannot be controlled by medications ( > 150/100 mmHg despite optimal medical therapy)
* History of HIV infection
* Active clinically serious infections ( > grade 2 NCI-CTC version 3.0)
* Known Central Nervous System tumors including metastatic brain disease
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Active disseminated intravascular coagulation, or patients prone to thromboembolism
* Patients undergoing renal dialysis
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehler, MD, Principal Investigator — Johannes Gutenberg University Mainz, I. Med. Klinik
Locations (11):
- Germany (11):
  - Klinikum der Johannes Gutenberg-Universität Mainz, I. Med. Klinik, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Jena, Klinik für Innere Medizin, Innere Medizin II, D-07740 Jena
  - Universitätsklinikum Hamburg-Eppendorf, I. Med. Klinik, Zentrum für Innere Medizin, Martinistr. 3, D-20248 Hamburg
  - Klinikum Fulda gAG, Tumorklinik, Pacelliallee 4, D-36043 Fulda
  - Klinikum der Johann-Wolfgang Goethe-Universität, Innere Medizin I, Theodor-Stern-Kai 7, D-60590 Frankfurt
  - Universitätsklinikum des Saarlandes, Klinik für Innere Medizin II, Kirrberger Str., Gebäude 41, D-66421 Homburg/Saar
  - Klinikum der Universität München, Medizinische Klinik II, Marchioninistr. 15, D-81377 München
  - Klinikum rechts der Isar, TU München, II. Medizinische Klinik und Poliklinik, Ismaningerstr. 22, D-81675 München
  - II. Med. Klinik, Leopoldina-Krankenhaus der Stadt Schweinfurt, Gustav-Adolf-Str. 8, D-97422 Schweinfurt
  - Klinikum Esslingen, Esslingen am Neckar
  - Universitätsklinikum Halle, Innere Medizin I, Halle

REFERENCES:
- [Derived] Kaps L, Genc MA, Moehler M, Grabbe S, Schattenberg JM, Schuppan D, Pedersen RS, Karsdal MA, Mildenberger P, Maderer A, Willumsen N. Collagen turnover biomarkers to predict outcome of patients with biliary cancer. BMC Gastroenterol. 2025 Feb 4;25(1):53. doi: 10.1186/s12876-025-03645-0. PMID 39905306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in was on 27MAY2008 Last patient out was on 20JUL2011
Pre-assignment Details: Six patients were enrolled but never treated. 97 patients were treated with study drug.
Groups:
- Gemcitabine + Sorafenib: Gemcitabine + Sorafenib
  Sorafenib : Sorafenib 400 mg bid orally continuously
  Gemcitabine : Gemcitabine 1000 mg/m2 body surface i.v. first cycle at day 1, 8, 15, 22, 29, 36, 43. Next cycles at day 1, 8, 15.
- Gemcitabine + Placebo: Gemcitabine + Placebo
  Gemcitabine : Gemcitabine 1000 mg/m2 body surface i.v. first cycle at day 1, 8, 15, 22, 29, 36, 43. Next cycles at day 1, 8, 15.
  Placebo : Placebo
Period: Overall Study
Arm/Group | Gemcitabine + Sorafenib | Gemcitabine + Placebo
Started | 49 | 48
Completed | 9 | 6
Not Completed | 40 | 42
Not completed — Death | 37 | 33
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other reason | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine + Sorafenib | Gemcitabine + Placebo | Total
Number analyzed (Participants) | 49 | 48 | 97
Age Continuous [Mean (Standard Deviation); unit: years] | 62.59 (9.01) | 63.23 (11.92) | 62.91 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 29 | 25 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 49 | 48 | 97
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 49 | 48 | 97
Type of Adenocarcinoma [Number; unit: participants]
  Adeno carcinoma, gall bladder | 6 | 7 | 13
  Adeno carcinoma, intrahepatic bile ducts | 33 | 29 | 62
  Adeno carcinoma, hepatic metastases | 10 | 12 | 22
Grading of adenocarcinoma [Number; unit: participants]
  1 (well differentiated) | 2 | 0 | 2
  2 (moderately differentiated) | 23 | 30 | 53
  3 (poorly differentiated) | 20 | 13 | 33
  4 (undifferentiated) | 1 | 0 | 1
  Missing | 3 | 5 | 8
Time since histological diagnosis [Mean (Standard Deviation); unit: days] — is defined as difference between date of first histological diagnosis and date of first visit
  days | 158.86 (347.69) | 275.81 (748.51) | 216.73 (581.55)
ECOG Performance Status [Number; unit: participants]
  0 | 30 | 35 | 65
  1 | 17 | 8 | 25
  2 | 0 | 1 | 1
  3 | 0 | 0 | 0
  4 | 0 | 0 | 0
  Missing | 2 | 4 | 6
Number of target lesions [Number; unit: participants]
  1 | 18 | 17 | 35
  2 | 16 | 10 | 26
  3 | 4 | 9 | 13
  4 | 4 | 4 | 8
  5 | 4 | 7 | 11
  6 | 1 | 1 | 2
  7 | 2 | 0 | 2
Number of non-target lesions [Number; unit: participants]
  1 | 23 | 16 | 39
  2 | 6 | 16 | 22
  3 | 6 | 8 | 14
  4 | 2 | 0 | 2
  5 | 1 | 0 | 1
  Missing | 11 | 8 | 19
Sum Sizes of target lesions [Mean (Standard Deviation); unit: mm] | 89.17 (56.29) | 95.02 (54.07) | 92.06 (54.07)

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The primary endpoint is the progression-free survival (PFS) defined as the time from start of treatment to first documentation of objective tumor progression or to death due to any cause, whichever occurs first during treatment or follow-up period. For patients not known to have died as of the data cut-off date and who do not have objective progressive disease, PFS will be censored at the date of the last objective progression-free disease assessment. For patients who receive subsequent anticancer therapy (after discontinuation from the study drug) prior to objectively determined disease progression or death, PFS will be censored at the date of the last objective progression-free disease assessment prior to post-discontinuation anti-cancer therapy. Acceptable documentation of objective disease progression status consists of objective assessments using CT scan assessment method.
Time Frame: one year
Population: All subjects who receive at least one dose of trial treatment are included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gemcitabine + Sorafenib | Gemcitabine + Placebo
Number analyzed (Participants) | 49 | 48
days | 91 [54 to 218] | 148 [105 to 233]
Statistical Analysis 1: Comparison: Gemcitabine + Sorafenib vs Gemcitabine + Placebo; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.281, 95% CI 2-sided [0.811 to 2.023]

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is measured from start of treatment to death due to any cause until end of follow-up period. Time to last observation will be used if a patient has not died and OS for the patient will be considered censored at the date of the last observation.
Time Frame: one year
Population: All subjects who receive at least one dose of trial treatment are included in the analysis
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gemcitabine + Sorafenib | Gemcitabine + Placebo
Number analyzed (Participants) | 49 | 48
days | 255 [166 to 384] | 341 [306 to 488]
Statistical Analysis 1: Comparison: Gemcitabine + Sorafenib vs Gemcitabine + Placebo; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.747 to 1.927]

3. Secondary Outcome: Best Overall Response
Description: Best Overall Response (BOR) is defined as the best tumor response (confirmed partial or complete response, stable disease) that is achieved during treatment or within 30 days after termination of active therapy that is confirmed according to the RECIST tumor response criteria. Best response is determined from the sequence of responses assessed. For complete response (CR) or partial response (PR), best response must be confirmed by a second assessment within 4 -6 weeks.
  Two objective status determinations of CR before progression are required for a best response of CR.
  Two determinations of PR or better before progression, but not qualifying for a CR, are required for a best response of PR.
  Best response of Stable Disease (SD) is defined as disease that does not meet the criteria of CR, PR or Progressive Disease (PD) and has been evaluated at least one time, at least 6 weeks after baseline assessment.
Time Frame: one year
Population: All subjects who receive at least one dose of trial treatment are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Sorafenib | Gemcitabine + Placebo
Number analyzed (Participants) | 49 | 48
participants
  Complete response | 0 | 0
  Partial response | 4 | 3
  Stable disease | 24 | 27
  Progressive disease | 0 | 0
  Missing | 21 | 18

4. Secondary Outcome: Time to Objective Response
Description: Time to Objective Response (OR) is defined as the time from start of treatment to objective tumor response (CR or PR) is first documented according to the RECIST tumor response criteria during treatment or until 30 days after termination of active therapy. Response must subsequently be confirmed. For subjects failing to achieve an objective response and who did not progress during the trial, time to objective response will be censored at their last date of tumor evaluation.
Time Frame: one year
Population: All subjects who receive at least one dose of trial treatment and had no progression during the trial are included in the analysis
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Gemcitabine + Sorafenib | Gemcitabine + Placebo
Number analyzed (Participants) | 24 | 25
days | NA [NA to NA] — it was not possible to calculate the median due to high number of censored observations | NA [NA to NA] — it was not possible to calculate the median due to high number of censored observations

ADVERSE EVENTS:
Arm/Group | Gemcitabine + Sorafenib | Gemcitabine + Placebo
Serious Adverse Events (participants affected / at risk) | 33/49 | 35/48
Other Adverse Events (participants affected / at risk) | 47/49 | 46/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Sorafenib (N=49) | Gemcitabine + Placebo (N=48)
Fever (General disorders) | 6 (8) | 5 (6)
General physical health deterioration (General disorders) | 6 (9) | 6 (6)
Pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Bile duct stent insertion (Surgical and medical procedures) | 1 (2) | 0 (0)
Biliary drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cholangitis suppurative (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (3) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 7 (7) | 3 (4)
Cholestasis (Hepatobiliary disorders) | 4 (4) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Sorafenib (N=49) | Gemcitabine + Placebo (N=48)
Fatigue (General disorders) | 26 (32) | 28 (32)
Pyrexia (General disorders) | 11 (17) | 15 (26)
General physical health deterioration (General disorders) | 0 (0) | 5 (6)
Oedema peripheral (General disorders) | 4 (4) | 11 (14)
Influenza like illness (General disorders) | 4 (4) | 3 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 16 (17) | 10 (10)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 5 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15 (19) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 11 (13) | 15 (15)
Leukopenia (Blood and lymphatic system disorders) | 15 (22) | 16 (23)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 4 (6) | 7 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (79) | 23 (45)
Abdominal pain (Gastrointestinal disorders) | 8 (11) | 4 (4)
Ascites (Gastrointestinal disorders) | 2 (2) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 17 (24) | 13 (13)
Vomiting (Gastrointestinal disorders) | 10 (11) | 10 (16)
Oral disorder (Gastrointestinal disorders) | 10 (11) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 4 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (11) | 11 (12)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9) | 9 (14)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (15) | 25 (31)
Headache (Nervous system disorders) | 3 (3) | 5 (6)
Paraesthesia (Nervous system disorders) | 8 (9) | 6 (6)
Polyneuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 8 (9)
Hypertension (Vascular disorders) | 5 (7) | 3 (3)
Hypertensive crisis (Vascular disorders) | 3 (4) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (9) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 11 (13) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Weight decreased (Investigations) | 12 (12) | 5 (5)
Haemoglobin decreased (Investigations) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Sleep disorder (Psychiatric disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes